CLINICAL TRIAL: NCT01965457
Title: Assessment of Adenoidal Obstruction in Children : Clinical Signs Versus Flexible Nasal Endoscopy and Roentgenographic Findings
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ohad Ronen, Senior Physician, Carmel Medical Center
Other Study IDs: AdeQ
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Obstructive Sleep Apnea; Nasal Obstruction
Keywords: obstructive sleep apnea; pediatric; adenoid hypertrophy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The term adenoids describes lymphoid tissue on the superior and posterior walls of the nasopharynx, and their hypertrophy is a common condition of childhood. When enlarged, adenoids can obstruct the nasopharyngeal airway and cause mouth-breathing, hyponasal voice, and snoring. In more severe cases, obstructive sleep apnea (OSA) may result, which carries potential risk of neurocognitive disturbance, growth failure, and heart-lungs disease. Adenoid hypertrophy can also be associated with otitis media with effusion, possibly through Eustachian tube dysfunction or chronic adenoidal infection.

Methods for identification of adenoid hypertrophy include the clinical history, examination, imaging (eg, plain lateral x-ray), or by nasal endoscopy witch enable direct visualization of the nasal cavity with dynamic evaluation of any nasal airway obstruction.

Objectives :

The aim of this study is to prospectively examine invasive and non-invasive office procedures to assess adenoids hypertrophy, including clinical history, x-ray imaging, and nasal endoscopy.

Methods :

Prospective, observational study in pediatric patients aged 2-18 that will be referred to the otolaryngology pediatric 'Clalit' clinic in Haifa after x-ray imaging and an informed consent.

1. Nasal Obstruction Index (NOI) The NOI questionnaire for history and physical exam will be evaluated at the clinic, as described by Paradise grading system.
2. Plain lateral x-rays Plain lateral X-rays of the patients will be evaluated only if the patients had them at the time of referral. Adenoidal obstruction will be assessed by Fujioka's Adenoid-Nasopharynx ratio.
3. Fiberoptic nasal endoscopy (FNE) Fiberoptic analysis will be done as an office procedure using a 2.4mm Storz nasal flexible endoscope following an application of Lidocaine gel locally into the nostril and on the endoscope distal end. Adenoidal obstruction will be assessed by Parikh grading system.

ELIGIBILITY:
Inclusion Criteria:

* age 2-18
* performed lateral cervical radiograph
* nasal obstruction
* signed informed consent by caregiver

Exclusion Criteria:

* previous adenoidectomy
* recent upper airway infection
* anatomic anomaly
* allergic rhinitis
* known obstructive sleep apnea

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 2-18 with suspected adenoid hypertrophy
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Adenoid Size Assessment | baseline
  Adenoid size assessment through a questionaire, physical exam, fiberoptic examination and lateral cervical radiographs.

SECONDARY OUTCOMES:
Efficacy of lateral cervical radiographs and fiberoptic exams | baseline
  A measurement of cases that the exam was not possible to perform or was not in good quality will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Cohen-Kerem, Md, Principal Investigator — Carmel Medical Center, Haifa
Locations (1):
- Armon Clinic, Haifa, Israel